CLINICAL TRIAL: NCT00367757
Title: Open, Prospective, Randomized Trial Comparing Trigger vs Substrate vs Hybrid Approaches for AF Ablation
Brief Title: STAR-AF:Substrate Versus Trigger Ablation for Reduction of Atrial Fibrillation Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AF06002AF
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation
Keywords: paroxysmal atrial fibrillation; persistent atrial fibrillation; high burden of atrial fibrillation; atrial fibrillation ablation; Pulmonary vein isolation; AF trigger; complex fractionated electrograms; CFE; CFAE; complex fractionated atrial electrograms; refractory antiarrhythmic medication; PVAI; Ensite NavX; NavX; CoolPath catheter; irrigated ablation catheter; high burden of paroxysmal or persistent atrial fibrillation; candidates for AF ablation; symptomatic AF; AF is refractory to at least one antiarrhythmic medication
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PVI group (Other): Trigger-based ablation guided by pulmonary vein antrum isolation
  Interventions: Procedure: Ablate AF triggers via PVI
- CFAE group (Other): Substrate-based ablation using an approach targeting CFAEs
  Interventions: Procedure: Substrate via CFAEs
- Combined group (Other): Combined trigger and substrate based approach
  Interventions: Procedure: Combined approach for AF ablation

INTERVENTIONS:
Procedure: Ablate AF triggers via PVI — Trigger-based ablation guided by pulmonary vein antrum isolation
  Arms: PVI group
Procedure: Substrate via CFAEs — Substrate-based ablation using an approach targeting CFAEs
  Arms: CFAE group
Procedure: Combined approach for AF ablation — Combined trigger and substrate based approach
  Arms: Combined group

SUMMARY:
Patient Population: Patients with AF that is symptomatic and refractory to at least one antiarrhythmic medication. Patients must have AF that is paroxysmal (>4 episodes within 6 months, two episodes >6 hours within 1 year) or persistent (sustained episode <6 months terminated by cardioversion or drug).

Purpose: To compare a trigger-based technique (pulmonary vein isolation) to a substrate-based technique (high-frequency, fractionated EGMs) to a combined approach for AF ablation

DETAILED DESCRIPTION:
Interventions: Patients will be randomized to either wide circumferential pulmonary vein isolation ("trigger") or ablation of high-frequency, fractionated electrograms during AF ("substrate"), or a hybrid approach combining trigger and substrate. Both techniques will be performed with NavX mapping system and a standardized ablation catheter. Endpoint of PVI will be isolation of all four PVs documented by circular catheter. Endpoint for substrate-based ablation will be termination and noninducibility of AF. Up to 2 procedures will be allowed within 6 months. A 2 month blanking period will be allowed after each procedure during which early recurrences will not be counted.

Outcomes:

* Recurrence of atrial fibrillation or other atrial tachycardia at 3, 6, and 12 months post-initial procedure.
* Recurrence will be defined by symptoms and/or ECG/Holter data showing AF > 2 mins
* Occurrence of adverse events in each group post-procedure.
* Quality of life assessment at 6 and 12 months post-initial procedure.

Followup:

* 3, 6, and 12 months post-initial procedure.
* Clinical data, ECG, Holter, loop recorder at baseline and at each visit.
* QOL at baseline, 3, 6 and 12 months post-initial procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 or greater.
* "high burden" of paroxysmal atrial fibrillation or persistent atrial fibrillation
* candidates for AF ablation based on AF that is symptomatic and refractory to at least one antiarrhythmic medication.
* At least one episode of AF must have been documented by ECG or Holter within 12 months of randomization in the trial.
* continuous anticoagulation with warfarin (INR 2-3) for >4 weeks prior to the ablation.
* Patients must be able and willing to provide written informed consent to participate in the clinical trial.

Exclusion Criteria:

* chronic atrial fibrillation.
* Patients with AF felt to be secondary to an obvious reversible cause.
* inadequate anticoagulation as defined in the inclusion criteria.
* left atrial thrombus or spontaneous echo contrast on TEE prior to procedure.
* contraindications to systemic anticoagulation with heparin or coumadin.
* previously undergone atrial fibrillation ablation.
* left atrial size > 55 mm.
* Patients who are or may potentially be pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2006-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation at 3 months post-first ablation procedure off antiarrhythmic medications. | 3 months
Freedom from atrial fibrillation at 6 and 12 months post-first ablation procedure off antiarrhythmic medications. | 12 months

SECONDARY OUTCOMES:
Freedom from atrial fibrillation on or off antiarrhythmic medications at 3, 6 and 12 months post-first ablation procedure. | 12 months
Freedom from atrial fibrillation and other atrial arrhythmias at 3, 6 and 12 months post-first ablation procedure. | 12 months
Incidence of peri-procedural complications including stroke, PV stenosis, cardiac perforation, esophageal injury, and death. | 12 months
Procedure duration at ablation. | At intervention
Fluoroscopy time at ablation. | At intervention
Quality of life measurements (SF-36) at baseline, 3, 6 and 12 months post-first procedure. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Atul Verma, Dr., Principal Investigator — Southlake Regional health Center
Locations (8):
- Canada (4):
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Montreal Heaert Institute, Montreal, Quebec
  - McMaster University, Hamilton
  - Victoria Cardiac Arrhythmia Trials Inc - Royal Jubilee, Victoria
- Italy (2):
  - Clinica Santa Maria, Bari, Apulia
  - Ospedale Regionale Ca'Foncello, Treviso
- Haukeland Universitetssykehus, Bergen, Haukeland, Norway
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

REFERENCES:
- [Derived] Verma A, Mantovan R, Macle L, De Martino G, Chen J, Morillo CA, Novak P, Calzolari V, Guerra PG, Nair G, Torrecilla EG, Khaykin Y. Substrate and Trigger Ablation for Reduction of Atrial Fibrillation (STAR AF): a randomized, multicentre, international trial. Eur Heart J. 2010 Jun;31(11):1344-56. doi: 10.1093/eurheartj/ehq041. Epub 2010 Mar 9. PMID 20215126